CLINICAL TRIAL: NCT05579483
Title: Prediction of Dietary Intervention Efficacy in Mild Ulcerative Colitis Patients Based on Fecal Microbiome Signatures
Acronym: PREDUCTOME
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wageningen University (Other)
Collaborators: Winclove Probiotics B.V. (Industry); China Scholarship Council (Unknown)
Responsible Party: Principal Investigator, Erwin Zoetendal, Associate professor, Wageningen University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NL79442.091.22; NL79442.091.22 (Other: METC Oost Nederlands)
Record Dates: First submitted 2022-10-04; First posted 2022-10-13 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Ulcerative Colitis
Keywords: prebiotics; ulcerative colitis; gut microbiome signature; fiber intake; prediction
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Prebiotics

STUDY DESIGN:
Intervention Model Description: A randomized, placebo-controlled, parallel, double-blind trial with two intervention arms and two control (placebo) arms.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Neither the investigator, the participants, nor the outcome assessor will know who received what. No Care Provider is included in this trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Predicted responders with prebiotics (Experimental): Predicted responders, which are defined as UC patients having a relative abundance of Bacteroidetes <=10% in their feces, will receive 6 grams of prebiotics per day.
  Interventions: Dietary Supplement: Prebiotics
- Predicted responders with placebo (Placebo Comparator): Predicted responders, which are defined as UC patients having a relative abundance of Bacteroidetes <=10% in their feces, will receive 6 grams of placebo per day.
  Interventions: Dietary Supplement: Placebo
- Predicted non-responders with prebiotics (Experimental): Predicted non-responders, which are defined as UC patients having a relative abundance of Bacteroidetes >=15% in their feces, will receive 6 grams of prebiotics per day.
  Interventions: Dietary Supplement: Prebiotics
- Predicted non-responders with placebo (Placebo Comparator): Predicted non-responders, which are defined as UC patients having a relative abundance of Bacteroidetes >=15% in their feces, will receive 6 grams of placebo per day.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Prebiotics — The prebiotics consists of three non-digestible carbohydrates (40% acacia gum, 20% partially hydrolyzed guar gum, and 40% resistant starch). During the 8-week intervention, two sachets (3 g per sachet) will be consumed per day, one in the morning and one in the evening.
  Arms: Predicted non-responders with prebiotics; Predicted responders with prebiotics
Dietary Supplement: Placebo — The placebo consists of two digestible carbohydrates (20% maltodextrin and 80% corn starch). During the 8-week intervention, two sachets (3 g per sachet) will be consumed per day, one in the morning and one in the evening.
  Arms: Predicted non-responders with placebo; Predicted responders with placebo

SUMMARY:
A double-blind randomized placebo-controlled parallel trial with two intervention arms and two placebo arms and a period of eight intervention weeks to validate the prediction that prebiotics could induce a higher response in mild UC patients with certain fecal microbiome signatures.

DETAILED DESCRIPTION:
Rationale: Ulcerative colitis (UC) patients respond differently to treatments/interventions (e.g. diet/fecal microbiota transplantation), but the reason for this individual specificity remains unknown. The investigators hypothesize that the baseline fecal microbiota composition determines the efficacy of a treatment/intervention, and potential responders, i.e. patients showing symptoms improvement after treatment, can be predicted based on fecal microbiota composition.

Objective: The primary objective is to validate the prediction that prebiotics intervention boosts butyrate production and thereby induces a higher response (lower mean Patient Simple Clinical Colitis Activity Index (P-SCCAI) score) in mild UC patients with low intestinal Bacteroidetes levels (predicted responders), but not in those with high intestinal Bacteroidetes levels (predicted non-responders) at T = 8 weeks. The secondary objectives are to study the effects of prebiotics intervention on disease activity over time (T = 0, 4, 8, 12 and 60 weeks), mucosal inflammation, gastro-intestinal (GI) complaints, stool consistency, stool frequency, fecal microbiota composition, fecal short-chain fatty acids concentrations, quality of life, number of participants with increased or decreased medication use, and incidence of adverse events in mild UC patients.

Study design: This study is a four-arm double-blind randomized placebo-controlled parallel trial. It consists of a screening stage in which mild UC patients will be assigned to be predicted responders or predicted non-responders based on fecal Bacteroidetes levels. Afterwards the predicted responders and non-responders will be assigned to either the prebiotics group (arm 1 and 3) or placebo group (arm 2 and 4).

Study population: Adult subjects aged 18-65 years and body mass index 18-30 kg/m2 with mild UC defined by P-SCCAI (3-5 points in a 19-point scale), with at least one relapse in the last two years.

Intervention: An 8-week intervention period with four parallel arms: 1) predicted responders with prebiotics treatment (acacia gum, partially hydrolyzed guar gum, and resistant starch), 2) predicted responders with placebo (maltodextrin and corn starch), 3) predicted non-responders with prebiotics treatment, 4) predicted non-responders with placebo, during which the study participants consume the respective supplement (3 grams, twice daily).

Main study parameters/endpoints: The main parameter is the response (mean P-SCCAI score) between arms at T = 8 weeks. The secondary parameters are the disease activity over time at T = 0, 4, 8, 12, and 60 weeks, mucosal inflammation (fecal calprotectin), gastro-intestinal (GI) complaints, stool consistency, stool frequency, fecal microbiota composition, fecal short-chain fatty acids concentrations, health-related quality of life, number of participants with increased or decreased medication use, and incidence of adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects aged 18 to 65 years
2. Body Mass Index (BMI) between 18 and 30 kg/m2 (self-reported)
3. Ulcerative Colitis confirmed via previous endoscopy and histology
4. Mild active UC as defined by P-SCCAI score of 3 to 5 (range 0 to 19)
5. Frequent relapse (at least one exacerbation in the last two years)
6. No known allergy to any components of the study product (self-reported)
7. Signed informed consent
8. Stable UC medication defined as no switch to other medication or no dose change
9. Mobile phone on which apps (used for questionnaires) can be downloaded (iOS version 9 and newer, Android version 4.4 and newer. Phones manufactured after 2013 are usually suitable)
10. Stable dietary pattern during the study

Exclusion Criteria:

1. Any other underlying disease of the GI-tract or previous bowel surgery, except cholecystectomy and appendectomy
2. Pregnancy or intending to become pregnant during the study
3. Use of medication that can interfere with the study outcomes, as judged by the medical supervisor
4. The need for antibiotic use during the intervention period
5. Systemic antibiotics and proton pump inhibitors (except for omeprazole and pantoprazole with dosage <20 mg), prebiotic supplements, probiotic supplements four weeks prior to study start
6. Currently participating in another intervention study
7. Acquaintances of anyone in the research team

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Response between arms at T = 8 weeks | Response at the end the intervention (T= 8 weeks)
  Within each arm, response will be determined by the mean Patient Simple Clinical Colitis Activity Index (P-SCAAI) score on a nineteen-point scale (from "0: no symptoms" to "19: severest symptom"). It refers to disease activity during the previous week, with higher scores representing worse disease symptoms.

SECONDARY OUTCOMES:
Disease activity over time (T= 0, 4, 8, 12, and 60 weeks) | Disease activity during and after the intervention (at T= 0, 4, 8, 12, and 60 weeks)
  Disease activity will be determined by the Patient Simple Clinical Colitis Activity Index (P-SCAAI) score on a nineteen-point scale (from "0: no symptoms" to "19: severest symptom"). With P-SCCAI score <= 2 being regarded as clinical remission, and a decrease in the P-SCCAI score by more than two points from baseline being regarded as clinical response. Comparisons will be made between groups as well as within subjects over time.
Mucosal inflammation | Change during and after the intervention (at T= 0, 8, 12, and 60 weeks)
  Mucosal inflammation will be determined by the fecal calprotectin level, which is a biomarker of inflammation and disease activity.
GI complaints | Change during the intervention (at T= 0, 4, and 8 weeks)
  The GI complaints will be assessed by the (gastrointestinal symptom rating scale) GSRS questionnaire, which has a seven-point graded scale where 1 represents the absence of troublesome symptoms and 7 represents very troublesome symptoms.
Stool consistency | Change during the intervention (at T= 0, 4, and 8 weeks)
  Stool consistency will be measured using the Bristol Stool Form Scale (7-point scale from 1=hard to 7=diarrhea) on a daily basis for 7 days
Stool frequency | Change during the intervention (at T= 0, 4, and 8 weeks)]
  Stool frequency will be measured by counting number of defecation on a daily basis for 7 days.
Fecal microbiota composition | Change during and after the intervention (at T= 0, 8, 12, and 60 weeks)
  Fecal microbiota composition will be determined by 16S rRNA gene sequencing.
Fecal short-chain fatty acids concentrations | Change during and after the intervention (at T= 0, 8, 12, and 60 weeks)
  Fecal short-chain fatty acids concentrations will be determined by HPLC.
Health-related quality of life | Change during the intervention (at T= 0, 4, and 8 weeks)
  Health-related quality of life will be assessed by short inflammatory bowel disease questionnaire (SIBDQ) with a seven-point graded scale where 1 represents very troublesome symptoms and 7 represents the absence of troublesome symptoms.
Number of participants with increased or decreased medication use | Change during and after the intervention (at T= 0, 4, 8, 12, and 60 weeks)
  It consists of the current medication use (e.g., aminosalicylates, corticosteroids, immunosuppressive agents, antimicrobial agents, and inhibitors of tumour necrosis factor-alpha (TNF- α)) with a downgrade meaning improvement and an upgrade meaning worsening of UC.
Incidence of adverse events | Change during the intervention (at T= 0, 4, and 8 weeks)
  Incidence of adverse events will be monitored by patient record and diary, these include all relapse-relevant information, including the need for systemic steroids, hospitalization, and surgery.

OTHER OUTCOMES:
Habitual dietary intake | FFQ will be taken at T= 0 (baseline).
  Habitual dietary intake including energy, nutrient, and fiber intake of the last month will be assessed by a validated food frequency questionnaire (FFQ) via FFQ-tool, a web-based interface tool.
Participants demographics and characteristics | This information will be collected at T= 0 (baseline).
  General information (e.g., sex, age, BMI, disease duration, age at diagnosis, smoking habit, UC location, type of treatment) will be collected

CONTACTS AND LOCATIONS:
Overall Officials: Erwin G Zoetendal, PhD, Principal Investigator — Laboratory of Microbiology, Wageningen University
Locations (1):
- Wageningen University, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No
As the data contains sensitive personal information researchers interested in the data can contact the principal investigator.

REFERENCES:
- [Background] Liu Z, de Vries B, Gerritsen J, Smidt H, Zoetendal EG. Microbiome-based stratification to guide dietary interventions to improve human health. Nutr Res. 2020 Oct;82:1-10. doi: 10.1016/j.nutres.2020.07.004. Epub 2020 Jul 21. PMID 32889252
- [Background] Fassarella M, Blaak EE, Penders J, Nauta A, Smidt H, Zoetendal EG. Gut microbiome stability and resilience: elucidating the response to perturbations in order to modulate gut health. Gut. 2021 Mar;70(3):595-605. doi: 10.1136/gutjnl-2020-321747. Epub 2020 Oct 13. PMID 33051190

DOCUMENTS (1):
  • Study Protocol (2022-07-26): https://cdn.clinicaltrials.gov/large-docs/83/NCT05579483/Prot_000.pdf